CLINICAL TRIAL: NCT05739669
Title: DigitalEPI - A Prospective Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding problems.
Sponsor: Karl Landsteiner Institute for Clinical Epilepsy Research and Cognitive Neurology (Other Government)
Collaborators: Brainhero GmbH (Industry); AIT Austrian Institute of Technology GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: DigitalEPI_Brainhero_CIP_002
Record Dates: First submitted 2023-01-23; First posted 2023-02-22 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: The EEG recordings will be gathered from each patient (single group) with two devices, in two different conditions and their quality assessed according to international standards by the IFCN.
  1. one EEG recording gathered with a CE-certified wet electrode device (Micromed Brain Quick; comparator device) by specialized staff in a clinician's office
  2. one EEG recording gathered with the investigational device "Atlas with dry electrodes" by specialized staff, in a clinician's office, immediately after (1)
  3. multiple EEG recordings gathered at home by non-specialized staff, for 14 days, using the investigational device "Atlas with dry electrodes" The study is exploratory.
  To further explore the diagnostic yield of recordings with the investigational device "Atlas with dry electrodes", the concordance of recorded dry electrode EEG data, semiautomatic analysis in encevis and data from the empatica EmbracePlus wrist device with established diagnoses will be investigated.
Masking Description: The quality of all the EEG recordings will be assessed by two highly qualified clinicians blinded to the recording condition and device. The diagnostic value of the home EEG monitoring will be evaluated by clinicians blinded to the patient's diagnosis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential EEG Recordings with a wet electrode device a dry electrode device in multiple settings (Other): * one recording per patient (epilepsy), performed by specialized staff in a clinic, with a CE-certified wet electrode EEG device (Micromed Brain Quick)
  * one recording per patient (epilepsy), performed by specialized staff in a clinic, with the investigational device "Atlas with dry electrodes"
  * multiple daily recordings from patients with epilepsy, gathered by lay people for 14 days, at home, with the investigational device "Atlas with dry electrodes"
  Interventions: Device: EEG recording with the comparator device Micromed Brain Quick; Device: EEG recording with the investigational device "Atlas with dry electrodes" clinic/specialized staff; Device: EEG recording with the investigational device "Atlas with dry electrodes" home/lay people

INTERVENTIONS:
Device: EEG recording with the comparator device Micromed Brain Quick — Each patient will undergo a visit in a clinic, during which a 15 minutes long EEG trace with a CE-certified wet electrode EEG Device (Micromed Brain Quick) will be recorded by specialized staff.
  Other Names: wet electrode EEG recording
Device: EEG recording with the investigational device "Atlas with dry electrodes" clinic/specialized staff — During the same visit when the wet electrode EEG is recorded, the patient will be subjected to a second 15 minutes long EEG recording with the investigational device "Atlas with dry electrodes", which will be conducted by specialized staff
  Other Names: dry electrode recording in a clinic, by specialists
Device: EEG recording with the investigational device "Atlas with dry electrodes" home/lay people — The patients will record their own EEGs at home daily for 14 days, using the investigational device "Atlas with dry electrodes"
  Other Names: dry electrode recording at home, by lay people / self-EEG recording at home

SUMMARY:
Not all patients with epilepsy requiring advanced checkups in specialized tertiary centers can be admitted for long-term video EEG monitoring. Home EEG recordings or home EEG monitoring using self-applicable EEG recording systems would therefore help overcome an unmet need in the treatment of such patients. Dry electrode EEG systems are more user-friendly than wet electrode EEG systems.

In this study, the quality of EEG recordings with a novel dry electrode EEG system (Atlas with dry electrodes) will be compared with the quality of recordings with a conventional wet electrode EEG system used in clinical practice. Secondly, the quality for medical reporting of self-recorded EEG at home by patients with the dry electrode EEG system (Atlas with dry electrodes) will be compared to recordings with the same system in a clinician's office by specialized staff. Thirdly, there will be an exploratory assessment of the value for diagnostics of EEG data from multiple home-recorded dry electrode EEGs, automatic analysis of those recordings and data from a wrist device.

The patients that fulfill inclusion criteria and do not meet exclusion criteria will all undergo the following:

* a visit to a clinic where a health care professional will record (1) their EEG activity for 15 minutes using a CE-certified EEG device with wet electrodes; and immediately after record (2) their EEG activity for 15 minutes using the investigational EEG device "Atlas with dry electrodes"
* self-record their EEG activity at home, using the EEG device "Atlas with dry electrodes", at least twice per day, for 14 days; during this phase, continuous non-invasive recordings of bio signals, i.e. heart rate, muscle activity, using the Empatica EmbracePlus device will be recorded and patients will report events or findings in a paper based study diary.
* a last visit to the clinic to return equipment, study diary and fill in questionnaires

DETAILED DESCRIPTION:
Background:

Advanced checkup of patients with epilepsy, especially in unclear or drug-resistant cases, includes a multiday inpatient hospital admission in specialized centers for long-term video and EEG recording. Not all patients can be admitted for such a prolonged period due to personal (familial) as well as professional obligations, comorbidities, or external factors such as limited healthcare resources in times of a global pandemic. Home EEG monitoring would enable clinicians to reach more patients requiring an advanced epilepsy checkup and save hospital resources.

Conventional EEG recording systems are intended to be used by specialized staff, e.g. EEG technicians, and are commonly based on wet electrodes that can't be self-applied. Brainhero GmbH has developed a portable wireless wet electrode EEG system that is CE certified as a medical product class IIa. This EEG system can easily be modified into a dry electrode system to be self-applied by patients.

EEG interpretation is time-consuming and requires a high degree of specialization. Automatic EEG analysis based on AI algorithms has proven to facilitate standardized EEG reporting and save resources.

Combining above considerations in a telehealth setting would allow for home-monitoring of patients with epilepsy.

Objectives and Hypoteses:

The study objectives are based on an explorative trial design. However, the investigators are interested in including the data gathered in this study in a further, larger-scale clinical trial. To this end, they outlined the null and alternative hypotheses based on a design estimated to be used at a larger scale. It is expected that the results will enable the refining of experimental design and appropriate sample size calculation for a consecutive trial.

Primary Objective: study feasibility

The study's primary objective is to evaluate the feasibility of the study design. The following outcomes will be evaluated:

* The percentage of high-quality recordings that can be gathered by specialized staff in clinical practice using the new dry electrode system
* The percentage of high-quality recordings that can be gathered at home by non-professional users using the new dry electrode system
* Whether 2 recordings per day for 14 days are sufficient to generate sufficient information to reach a diagnosis or not.
* The degree of compliance and adherence of the study participants to the study protocol
* Identification of characteristics (social, demographic, information from the electronic health records etc) of successful study participants

Secondary Objective: descriptive statistics The secondary objective of this study is to generate data relevant to the design of a further, larger scale clinical trial. To this end, three aims were outlined, each with individual hypotheses.

Primary exploratory aim

The primary exploratory aim of the study is to exploratively compare the quality of EEG recordings generated by a novel dry electrode EEG system with EEG recordings gathered with a conventional wet electrode EEG system used in clinical practice. The comparison will be based on visual assessment by two experienced clinical neurophysiologists and power spectrum analysis.

Hypotheses:

H1: There is no difference in quality for medical reporting between the dry electrode EEG and the conventional EEG when they are recorded in the clinician's office under the same conditions, by specialized staff.

H0: There is a difference in quality for medical reporting between the dry electrode EEG and the conventional EEG when they are recorded in the clinician's office under the same conditions, by specialized staff.

Rationale: Conventional EEG is the gold standard of quality for EEG recordings, whereas dry electrodes are expected to give a lower-quality signal and therefore result in a lower-quality recording.

Secondary exploratory aim

A further aim of the study is to exploratively compare the quality for medical reporting of self-recorded EEG at home by patients with the dry electrode EEG system with the quality of recordings with the same system at the study center by specialized staff. The comparison will be based on the visual assessment by two experienced clinical neurophysiologists and power spectrum analysis.

Hypotheses:

H1: There is no difference in quality for medical reporting between the dry electrode EEG recorded at home by the patient and the dry electrode EEG recorded in a clinician's office by specialized staff.

H0: There is a difference in quality for medical reporting between the dry electrode EEG recorded at home by the patient and the dry electrode EEG recorded in a clinician's office by specialized staff.

Rationale: It is expected that the specialized staff with significant experience in recording EEGs will be able to obtain a better-quality recording than the lay people that are just learning to do this and will record it without the supervision of the qualified experts.

Tertiary exploratory aim

The tertiary exploratory aim of the study refers to an exploratory analysis, where the investigators will assess the value for diagnostics of EEG data from multiple home-recorded dry electrode EEGs, automatic analysis of those recordings, and data from a wrist device.

The patients included in this study have a diagnosis based on several evaluations, including conventional EEG; this is called diagnosis A. The investigators will exclude the conventional EEG data from patient files of included patients and replace it with the dry electrode data and automatic analyses gathered in this pilot study, along with data recorded via a wrist device called Empatica EmbracePlus; based on the latter data the investigators will establish diagnosis B. The evaluators of diagnosis B will be blinded with respect to diagnosis A.

It is expected that the diagnosis based on EEG recordings obtained with dry electrodes, with most likely lower quality than the conventional EEGs, will not be as accurate as the diagnosis which relies on EEG recordings obtained with conventional EEG devices. However, given that the dry electrode EEGs recorded at home, when correctly performed, provide multiple time points and potentially more comprehensive medical information, the possibility that Diagnosis B is more comprehensive than diagnosis A. The validity of these assumptions will be explored as part of the tertiary exploratory objective in which the investigators aim to assess the concordance of diagnoses A and B.

Methods:

A minimum of 18 patients with a previously established diagnosis of epilepsy who are treated at the investigators' epilepsy clinics either in- or outpatient will be included in the study. Only patients who received a previous thorough diagnostic workup will be enrolled because no therapeutic intervention is planned in the present study. Because theinvestigators expect a drop-out rate of 20%, they will aim to recruit 18 patients to have 15 patients for analysis.

Possible study participants will be identified among all patients who attend a routine outpatient appointment or receive inpatient care including but not limited to VEM at the clinic that represents the clinical investigation site according to the inclusion criteria. Those patients will be approached by the study team, and informed about the study and the study information flyer as well as patient information will be handed out. After sufficient time for consideration and after giving informed consent patients will be enrolled.

1. Visit 1 - Instruction and supervised recording During a first study visit, all study procedures will be thoroughly explained, and patients will be instructed in using and self-applying the portable EEG-recording system, using the recording laptop, and using the Empatica E4 wristband.

   Before enrolling women of childbearing age, a pregnancy test will be conducted to exclude an unnoticed pregnancy. If any women of childbearing age should be enrolled in the study for more than one month, a monthly pregnancy test will be conducted. However, this is highly unlikely since study participation enrollment is 14 days.

   Both, an EEG with the routine clinical EEG system in use at the investigators' center (Micromed Brainquick wet electrode system) and an EEG with the portable EEG dry electrode system (Atlas EEG system with dry electrode cap) under the same conditions in the same room will be recorded sequentially following standards for digital EEG recordings by the IFCN [25].
2. Home recordings After visit 1, patients will start recording EEG at home twice daily in the morning and evening for 15 minutes for 14 days. Patients will be instructed to use the same room and surroundings for all recordings, remain seated in a quiet environment without disrupting external stimuli, and not use any other electronic devices such as smartphones, tablets, or smartwatches during the recordings. Additional recordings might be collected based on certain triggers. Those triggers include 1) known clustering of seizures at a certain time of the day, e.g. circadian clustering.

2) a feeling that an epileptic seizure might happen soon (= epileptic aura) 3) after an epileptic seizure Additionally, continuous non-invasive recordings of biosignals, i.e. heart rate, muscle activity, from Empatica EmbracePlus will take place and patients will report events or findings in a paper-based study diary.

The study team will be available to patients during office hours for questions or troubleshooting.

3. Final study visit After 14 days patients will take part in a final study visit at the investigation site where the equipment is returned and post-study questionaries will be filled out by patients.

Data collection and processing:

All data collected will be managed pseudonymized. Home EEG recordings will initially be saved locally to the recording laptop. Recordings will then be transferred ID-bound over the internet using the encrypted connection of Tresorit, which is accessible at the research workstation located at the investigators' center. Data from the Empatica EmbracePlus wristband device will be stored on the Empatica device and synced over Bluetooth via the Empatica App to the proprietary Empatica cloud service.

Further analysis will be performed after the patient returns the study equipment during the post study visit.

All recorded EEG files will be converted to DICOM for analysis based on scripts by Sigma Software Solutions OG and tracings will be visually inspected and an automatic and clinically validated analysis of IED and EEG trends will be performed in encevis on the research workstation with posthoc review of detected events by clinicians (=semiautomatic or hybrid approach). Data analysis will be done by KLI in collaboration with AIT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed epilepsy
* ≥ 1 seizure during the last year
* ≥ 1 routine EEG at the investigation center or VEM
* Age ≥ 18 years

Exclusion Criteria:

* History of PNES
* Inability to comply with the trial procedures
* Inability to give informed consent
* Pregnant and breastfeeding patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
% of good quality EEG recordings taken by specialised staff in a clinic with "Atlas with dry electrodes" | Initial visit in a clinic (one day)
  The routine wet-electrode EEG recorded during study visit 1 will be compared to the EEG recorded with the portable dry-electrode EEG system (investigational device). A visual analysis based on the percentage of artifact-contaminated EEG segments and the signal-to-noise ratios (according to IFCN standards) will be performed and recordings graded on a 1-3 numerical ordinal semi-quantitative scale:
  1. EEG is unrestrictedly usable for clinical reporting (i.e. the interpretation is not significantly compromised by technical artifacts, biological artifacts or any other technical aspect)
  2. EEG is limitedly usable for clinical reporting (i.e. the artifacts cause uncertainty with respect to diagnosis or therapy, but do not prevent the rater from deriving diagnostic findings)
  3. EEG is not usable for clinical reporting (i.e. a diagnostic finding could not be stated)
  The % of dry-electrode recordings scored with 1 or 2 (good quality) gathered by experts in the clinic will be reported.
% of good quality EEG recordings taken by lay people at home with "Atlas with dry electrodes" | 14 days, at home
  If visit 1 dry electrode EEG is rated as unrestrictedly usable for clinical reporting or limitedly usable for clinical reporting (grade 1 or 2 on the 1-3 scale outlined at Outcome 1), all dry electrode EEG home recordings will be again scored as listed in Outcome 1 (outcome measures 1, 2 or 3), and compared to visit 1 dry electrode EEG.
  The % of dry-electrode recordings scored with 1 or 2 (good quality) gathered at home by non-professional users using the new dry electrode system

SECONDARY OUTCOMES:
Number of participants that are diagnosed with epilepsy based on home recordings with "Atlas with dry electrodes" | 14 days, at home
  To explore the diagnostic yield of recordings with the dry electrode recording system, the concordance of recorded dry electrode EEG data, semiautomatic analysis in encevis and data from the empatica EmbracePlus E4 wrist device with established diagnoses will be investigated.
  The patients included in this study have a previously established diagnosis based on several evaluations, including conventional EEG; this is called Diagnosis A. The investigaros will exclude the conventional EEG data from patient files of included patients and replace it with the dry electrode data and automatic analyses gathered in this pilot study, along with data recorded via a wrist device called Empatica EmbracePlus; based on the latter data the investigators will establish diagnosis B. The raters of diagnosis B will be blinded with respect to diagnosis A.
  Concordance of diagnosis A with diagnosis B will be evaluated. The number of participants whose diagnosis B was epilepsy will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Baumgartner, MD, Principal Investigator — Department of Neurology, KLI Clinical Epilepsy Research - Clinic Hietzing, Vienna, Austria
Locations (1):
- Department of Neurology, Clinic Hietzing, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: No